CLINICAL TRIAL: NCT02060903
Title: A Randomized, Double-Blind, Multicenter, Vehicle-Controlled Study of the Efficacy and Safety of Abametapir Lotion 0.74% Administered for the Treatment of Head Lice Infestation
Brief Title: A Study of the Efficacy and Safety of Abametapir Lotion Administered for the Treatment of Head Lice Infestation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: Accelovance (Industry); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ha03-001
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Head Lice Infestation
Keywords: Head Lice; Hatchtech

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abametapir Lotion 0.74% w/w (Active Comparator): Single topical treatment administered to hair and scalp for 10 minutes. Applied at home by a subject/caregiver.
  Interventions: Drug: Abametapir Lotion 0.74% w/w
- Vehicle Lotion (Placebo Comparator): Single topical treatment administered to hair and scalp for 10 minutes. Applied at home by a subject/caregiver.
  Interventions: Drug: Vehicle Lotion

INTERVENTIONS:
Drug: Abametapir Lotion 0.74% w/w — Abametapir Lotion 0.74% was dispensed to subjects on Day 0 for self-administration at home on the same day.
  Other Names: Abametapir 0.74%
  Arms: Abametapir Lotion 0.74% w/w
Drug: Vehicle Lotion — Vehicle Lotion was dispensed to subjects on Day 0 for self-administration at home on the same day.
  Other Names: Vehicle
  Arms: Vehicle Lotion

SUMMARY:
The purpose of the study was to assess the efficacy, safety and tolerability of a single application of abametapir lotion 0.74% w/w compared to a vehicle control, when applied to the scalp and hair for 10 minutes at home.

DETAILED DESCRIPTION:
This was a randomized, double-blind, multicenter, vehicle-controlled, parallel-group study in subjects with active head lice infestation. The study was designed to assess the efficacy, safety and tolerability of a single application of abametapir lotion 0.74% w/w compared to a vehicle control, when applied to scalp and hair for 10 minutes at home.

Approximately 106 index subjects with their household members were enrolled into the study. A total of approximately 318 subjects were enrolled, assuming an average of 3 members per household participating in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged six months of age or older.
2. Is in good general health based on medical history.
3. Has active head lice infestation at Screening as determined by a trained evaluator with the exception of the male head of household who may self-assess as being lice-free. Active head lice infestation is defined as at least three live lice for the index subject and at least one live louse for the other household members.
4. The subject and/or their caregiver is physically able and willing to apply the Investigational Product at home.
5. Belongs to a household with an eligible index subject with active head lice infestation.
6. Agrees to an examination for head lice and to all visits and procedures throughout the study.
7. Has signed an informed consent and/or assent form.

Exclusion Criteria:

1. Had treatment (over-the-counter ), home remedy or prescription medication) for head lice within 14 days prior to Day 0.
2. Intends to use any other form of lice treatment from Day 0 through the Day 14 visit, unless provided as rescue therapy to this Protocol.
3. Intends to use a lice comb from the Day 0 through the Day 14 visit unless provided as rescue therapy to this Protocol.
4. Intends to cut their hair, use hair dye/bleach or have permanent wave hairstyling from Day 0 through the Day 14 visit.
5. Has a household member(s) who is infested with lice but is not willing or not eligible for enrollment.
6. Has a condition that, in the opinion of the Investigator, may increase the risk to the subject and/or the interpretation of the data.
7. Has visible skin/scalp condition(s) that are not attributable to head lice infestation, such as an erythema score that is >2, blisters, vesicles which, in the opinion of the investigative personnel or Sponsor, will interfere with safety and/or efficacy evaluations.
8. Has eczema or atopic dermatitis of skin/scalp.
9. Has had a prior reaction to Nix® or products containing permethrin.
10. Receiving systemic or topical medication, which in the opinion of the Investigator, may compromise the integrity of the safety and/or efficacy assessments.
11. Has received an investigational agent within 30 days prior to Day 0.
12. Does not have a known household affiliation with the household members (i.e., does not stay in one household consistently, or sleeps at one place for several nights and then at another place or location).

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sidgiddi, MD, Study Director — Dr. Reddy's Laboratories Inc.
Locations (7):
- United States (7):
  - Universal Biopharma Reserach INC, Dinuba, California
  - Axis Clinical Trials, Los Angeles, California
  - LSRN Reserach, West Palm Beach, Florida
  - Impact Clinical Trials, Las Vegas, Nevada
  - Haber Dermatology, Beachwood, Ohio
  - McKenzie Medical Center, McKenzie, Tennessee
  - Radiant reserach Inc., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Abametapir Lotion 0.74% w/w: Single topical treatment administered to hair and scalp for 10 minutes. Applied at home by a subject/caregiver.
  Abametapir Lotion 0.74% w/w
- Vehicle Lotion: Single topical treatment administered to hair and scalp for 10 minutes. Applied at home by a subject/caregiver.
  Vehicle Lotion
Period: Overall Study
Arm/Group | Abametapir Lotion 0.74% w/w | Vehicle Lotion
Started | 187 | 192
Completed | 183 | 185
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 0 | 7

BASELINE CHARACTERISTICS:
Population: The All Randomized Subjects population consisted of all subjects randomized into the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Abametapir Lotion 0.74% w/w | Vehicle Lotion | Total
Number analyzed (Participants) | 187 | 192 | 379
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.28 (12.11) | 16.58 (13.93) | 16.43 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 160 | 321
  Male | 26 | 32 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 142 | 162 | 304
  Not Hispanic or Latino | 45 | 30 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 181 | 191 | 372
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 187 | 192 | 379

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Index Subjects Who Are Lice-free at All Follow-up Visits Through to the Day 14 Visit.
Description: Proportion of index subjects randomized into the study who are lice free at all follow up visits through to the Day 14 visit. The index subject of a household was the youngest person within that household with at least 3 live lice present, as assessed over a period of up to 15 minutes at the Screening Visit.
Time Frame: 14 days
Population: The ITT population consisted of all 108 index subjects who were enrolled and randomized in the study.
Measure: Number; unit: participants
Arm/Group | Abametapir Lotion 0.74% w/w | Vehicle Lotion
Number analyzed (Participants) | 53 | 55
participants | 43 | 28

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from the start of treatment until 14 days following IP treatment (approximately 15 days).
Arm/Group | Abametapir Lotion 0.74% w/w | Vehicle Lotion
All-Cause Mortality (participants affected / at risk) | 0/186 | 0/188
Serious Adverse Events (participants affected / at risk) | 0/186 | 1/188
Other Adverse Events (participants affected / at risk) | 0/186 | 0/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abametapir Lotion 0.74% w/w (N=186) | Vehicle Lotion (N=188)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No